CLINICAL TRIAL: NCT04242251
Title: Novel Palliative Care Model for Advanced Cancer Patients: A Randomized Controlled Trial Study
Acronym: SPARKLE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/2963
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: Palliative Care; Cancer; Health Services Research
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person administering the patient reported outcome measures will be blinded to the participant's allocation to study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Management by primary oncologist. Referral to existing palliative care service initiated by primary oncologist if needed.
- SPARKLE intervention group (Experimental): Regular symptom monitoring and treatment of problems identified. Referral to existing palliative care services can also be initiated by the SPARKLE nurse if identified problems require follow up.
  Interventions: Other: SPARKLE Model of care

INTERVENTIONS:
Other: SPARKLE Model of care — Patients will receive the SPARKLE model of care in addition to usual oncologist-led care. The SPARKLE model will be led by a palliative medicine doctor and administered by nurses and staff without specific nursing or medical training. It utilizes a stepped care approach where all patients will initially have low-intensity model focused on weekly symptom monitoring through a patient-reported questionnaire. If any problems are identified, then patients step up to a higher-intensity care model where a nurse will conduct a phone assessment of the symptom problems. If the presence of symptoms is confirmed, patients step up again to an even higher-intensity care model where treatment of symptoms will be initiated by the SPARKLE nurse, depending on the severity of the problems. If the symptoms are not fully resolved, the patients will then step up to the highest-intensity care model which is an existing palliative care service- either palliative care outpatient clinic or home hospice.
  Arms: SPARKLE intervention group

SUMMARY:
This is a randomized controlled trial of the 'Supportive and Palliative care Review Kit in Locations Everywhere' (SPARKLE) intervention, an outpatient-based model of early palliative care. The SPARKLE intervention comprises regular symptom monitoring using questionnaires, early identification and prompt treatment of problems identified. Proactive screening for problems facilitates earlier palliative care interventions for advanced cancer patients, whenever needs arise.

DETAILED DESCRIPTION:
This is a randomized controlled trial to compare clinical outcomes between advanced cancer patients receiving and not receiving care from the SPARKLE care model, in addition to current oncologic-led palliative care model. The hypothesis is that the SPARKLE care model results in a) improved quality of life of both advanced cancer patients and their caregivers, and b) reduced acute healthcare utilization and costs by these patients.

Primary Study Aim: To determine the incremental effect of SPARKLE in addition to usual oncologist-led care on quality of life of advanced cancer patients. Patients' quality of life will be measured at baseline before randomization and 16 weeks after randomization using the Functional Assessment of Cancer Therapy - General (FACT-G).

Secondary Study Aim 1: To determine the incremental effect of SPARKLE in addition to usual oncologist-led care on caregivers' quality of life. Caregiver quality of life will be measured at baseline before randomization and 16 weeks after randomization using the Singapore Caregiver Quality of Life Scale (SCQOLS), which was validated among caregivers of advanced cancer patients in Singapore.17 The PI was part of the team, led by the applicant's mentor, that developed the SCQOLS.

Secondary Study Aim 2: To determine the effect of SPARKLE in addition to usual oncologist-led care on healthcare utilization and total healthcare costs, including the costs of delivering SPARKLE, from randomization until death. Healthcare utilization and cost data will be extracted from medical and billing data. SPARKLE costs will be captured prospectively using an Activity Based Costing Approach. The study hypothesis is that per capita healthcare costs will be lower in the SPARKLE model due to fewer admissions and shorter hospital lengths of stay when admitted.

A prospective randomized controlled trial design will be used to test the effectiveness of the SPARKLE model. The recruitment target is 240 patients with advanced cancers, defined as stage 4 solid tumors including lung, colorectal, nasopharyngeal and pancreatic cancers. Eligible participants are randomized to usual care or SPARKLE intervention group using randomized permuted blocks method generated by an independent statistician, with block size kept unknown to the clinical investigators/site personnel. A total of 240 caregivers will be recruited.

The study will take place in the National Cancer Centre of Singapore (NCCS).

ELIGIBILITY:
Patient participants Inclusion Criteria:

* Adult aged 21 and above
* Stage 4 solid tumor

Patient participants Exclusion Criteria:

* Unable to complete patient-reported outcome measures
* Already under the care of an existing palliative care service

Caregiver participants Inclusion Criteria:

- Adult aged 21 and above

Caregiver participants Exclusion Criteria:

* Unable to complete Singapore Caregiver Quality of Life Scale questionnaire
* Employed caregiver to patient participants

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy- General | 16 weeks
  Quality of life is scored on a scale of 0 to 108, with higher scores indicating better outcomes

SECONDARY OUTCOMES:
Singapore Caregiver Quality of Life Scale | 16 weeks
  Caregiver quality of life is scored on a scale of 0 to 100, with higher scores indicating better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Grace M Yang, MRCP, Principal Investigator — Consultant
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Yang GM, Ke Y, Ng XH, Neo PSH, Cheung YB. Proactive symptom monitoring to initiate timely palliative care for patients with advanced cancer: a randomized controlled trial. Support Care Cancer. 2025 Mar 5;33(3):249. doi: 10.1007/s00520-025-09311-1. PMID 40038129